CLINICAL TRIAL: NCT01046513
Title: PET Imaging of Nicotinic Acetylcholine Receptors With 2-[18F]F-A-85380-Injection, Initial Evaluation of Radiotracer in Human Volunteers
Brief Title: PET Imaging of Nicotinic Acetylcholine Receptors
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906364; 06-DA-N364
Record Dates: First submitted 2010-01-09; First posted 2010-01-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-28

CONDITIONS: Healthy Volunteers; Nicotine Dependence; Pharmacokinetics
Keywords: Nicotinic Acetylcholine Receptors; Neuroimaging; Positron Emission Tomography (PET); Alpha4beta2; Nicotine; Receptor Upregulation
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Central nicotinic acetylcholine receptors (nAChRs) are the primary target for the action of nicotine. In addition to being involved in tobacco dependence, they are also involved in a variety of brain disorders, including Alzheimer's and Parkinson's diseases. Researchers are interested in developing better ways to study the action of nAChRs to improve treatments for smoking cessation and other problems affected by these receptors. These new study methods may involve different radiotracers, which are drugs that can help show brain activity during positron emission tomography (PET) scanning.

Objectives:

- To evaluate the feasibility of using a radiotracer, 2-[18F]F-A-85380, in PET scanning of the brain.

Eligibility:

- Healthy volunteers between 21 and 45 years of age who do not use tobacco.

Design:

* Participants will be asked to avoid consuming alcohol or using a number of over-the-counter medications, including antihistamines, cough medicines, and nasal decongestants, for 5 days before the study day. Participants provide urine and breath samples at the start of the study to be tested for chemicals that may interfere with the study.
* Participants will visit the clinical center the morning of the day before the scanning session to provide blood and urine samples as required. Participants will return and be admitted for an overnight stay later that afternoon or evening.
* On the day of the study, participants will receive a single dose of the radiotracer 2-[18F]F-A-85380, and will have a series of PET scans over the next 7 hours and provide blood samples during that time. Participants will spend that night at the clinical center and leave on the morning after the end of the study.
* Participants will return for follow-up visits 2 weeks and 1 month after the end of the study.

DETAILED DESCRIPTION:
Background: Central nicotinic acetylcholine receptors (nAChRs) mediate a variety of brain functions and have been implicated in the pathophysiology of Alzheimer's and Parkinson's diseases, other CNS disorders (Tourette's syndrome, epilepsy, etc.), and nicotine dependence. These receptors are the primary target for the action of nicotine, which is believed to cause tobacco dependence. The availability of a suitable agent that could image nAChRs with PET in humans would allow scientists to monitor the nAChRs in vivo for the purpose of determining their roles in the pathogenesis of neurodegenerative diseases and nicotine dependence.

Scientific Goals: The immediate goal of the proposed study is to evaluate the feasibility of using a radiotracer, 2-[18F]F-A-85380, developed by scientists in the NIDA Brain Imaging Center for external imaging of nAChRs in the human brain.

Study Population: Healthy adult participants, males and females between 21 and 45 years of age, will be recruited for this study. The goal is to complete studies of 7 male and 7 female subjects.

Experimental Design and Method: After being medically cleared and giving informed consent, participants will receive a single dose of the radiotracer, 2 [18F]F A 85380-Injection, and will undergo a series of PET scans acquired over the next 7 hours after the injection. The PET scans will be used to determine the time course of the distribution of the injected radioactivity in those organs expected to receive the highest radiation exposure and in the brain.

Benefits to participants and/or society: This protocol will provide no direct benefits to the research participants other than routine medical screening and attention from the research staff. The knowledge gained in this study may lead to the availability of an agent for external monitoring of nAChRs using PET. This agent would be a valuable tool for determining the role of nAChRs in the pathogenesis of neuropsychiatric diseases, including nicotine dependence and for developing medications for diseases that respond to nicotinic agonists.

Risks to participants: There is some risk attendant to the PET scans in general, involving exposure to radiation, arterial catheterization and venous catheterization. In addition, there is risk related to the administration of this radiopharmaceutical, as it will be given to humans for the first time in this study. Medical supervision will be provided throughout the study. A plan for monitoring potential side effects of this radiotracer is given.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: Subjects will be male and female volunteers aged 21 to 45 years. All subjects must have a stable point of contact and must agree to return at 2 and 4 weeks after the PET study for laboratory screening and follow up evaluations.

EXCLUSION CRITERIA:

1. Psychiatric disease: DSM-IV criteria will be used (DSM-IV, APA, 1994). No subject with a current axis I diagnosis will be allowed. No subject with known claustrophobia will be allowed.
2. History of Drug Abuse: Volunteers reporting current or having a significant history of illicit drug abuse (single illicit substance use of more than 10 times in a lifetime for any given substance, except marijuana) will be excluded from the study. Volunteers reporting current use of nicotine will be excluded because nAChRs are usually elevated in smokers, and the purpose of this protocol is to determine the feasibility of measuring nAChRs in vivo. Including smokers at this time may provide results that are more variable and which may overestimate our ability to measure these receptors in nonsmokers. Subjects may use moderate amounts of alcohol and caffeine and smoke an occasional marijuana cigarette. Moderate alcohol use will be defined as less than ten drinks of liquor (1.5 oz) or the equivalent beer (12 oz) or wine (5 oz) per week. Moderate caffeine use will be defined as less than 500 mg of caffeine per day, where 100 mg is equivalent to 1 serving of coffee (5 oz serving), 2.5 servings (12 oz serving) of caffeinated soft drinks, or 2.5 servings of tea (5 oz serving). Occasional marijuana use will be defined as less than or equal to two marijuana cigarettes/month.
3. Current Medication Use: Volunteers may not currently use chronic (daily or for more than 10/14 days in the last month) prescription or over the counter medications, (including, but not limited to, anti-hypertensive, anti-allergy, pain). Over the counter or prescription medications may used on an occasional basis (for treatment of self-limited conditions, such as occasional headache, musculoskeletal discomfort, allergic symptoms or pain). All medications will be discontinued at least 5 days before the experimental session.
4. CNS disease: History of known structural brain abnormalities (e.g., neoplasm, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), history of head trauma (defined as documented loss of consciousness > 5 min or injury requiring hospitalization), history of seizures as an adult, sleep apnea.
5. Cardiovascular, pulmonary, or systemic disease: Repeated (measured on three separate occasions) diastolic blood pressure > 90 mm Hg, or systolic blood pressure > 150 mm Hg, known arrhythmia, symptomatic or known coronary artery disease; history of endocarditis, cerebral embolism, obstructive pulmonary disease, asthma, active tuberculosis, known endocrine disease (derangements in adrenal, thyroid, bone or reproductive function) known chronic renal or hepatic dysfunction, known HIV seropositive, known current autoimmune disease involving the CNS, type I diabetes mellitus, current gastrointestinal disease, gastritis or ulcers.
6. Special considerations for female subjects. Female participants who are currently pregnant or nursing will not be allowed to participate in this study. Female subjects will be given a serum pregnancy test (quantitative beta HCG) within 24 hours of each PET session.
7. Miscellaneous exclusionary criteria: Body mass index less than 20 or greater than 29. Hematocrit < 39.0 for males or < 35.0 for females.
8. Radiation exposure: Any subject who has participated in any research studies in which he/she received a radiation exposure that would result in combination with the present study, in a total effective radiation exposure (from research studies) exceeding 3.0 rem in a 13-week period or 5.0 rem in a year.
9. Novocain allergy.
10. Test of hand cubital artery patency for all subjects.
11. Women who are pregnant or lactating and children under the age of 21 will be excluded to avoid unnecessary exposure to radiation to these populations.
12. The presence within the body of metallic implants or materials that could be moved by the magnet of the MRI scanner: pacemakers, surgical implants, aneurysm clips, dental braces, bullet(s) or other metallic materials.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2007-08-31; Study Completion 2011-09-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Adler LE, Hoffer LJ, Griffith J, Waldo MC, Freedman R. Normalization by nicotine of deficient auditory sensory gating in the relatives of schizophrenics. Biol Psychiatry. 1992 Oct 1;32(7):607-16. doi: 10.1016/0006-3223(92)90073-9. PMID 1450287
- [Background] Bannon AW, Decker MW, Curzon P, Buckley MJ, Kim DJ, Radek RJ, Lynch JK, Wasicak JT, Lin NH, Arnold WH, Holladay MW, Williams M, Arneric SP. ABT-594 [(R)-5-(2-azetidinylmethoxy)-2-chloropyridine]: a novel, orally effective antinociceptive agent acting via neuronal nicotinic acetylcholine receptors: II. In vivo characterization. J Pharmacol Exp Ther. 1998 May;285(2):787-94. PMID 9580627
- [Background] Benwell ME, Balfour DJ, Anderson JM. Evidence that tobacco smoking increases the density of (-)-[3H]nicotine binding sites in human brain. J Neurochem. 1988 Apr;50(4):1243-7. doi: 10.1111/j.1471-4159.1988.tb10600.x. PMID 3346676